CLINICAL TRIAL: NCT05759754
Title: Treatment Effects of Traditional Chinese Medicine (Gu Shen Juan Yu Formula) in Children With Inherited Proteinuric Kidney Disease：A Multicenter, Open-Label, Two-Arm, Crossover Randomized Clinical Trial
Brief Title: Effects of Traditional Chinese Medicine (GSJYF) in Children With Inherited Proteinuric Kidney Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Fudan University (Other)
Collaborators: Anhui Provincial Children's Hospital (Other); Henan Provincial People's Hospital (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); Children's Hospital of Nanjing Medical University (Other); The Children's Hospital of Zhejiang University School of Medicine (Other); First Affiliated Hospital, Sun Yat-Sen University (Other); Shandong Provincial Hospital (Other Government); Xuzhou Children Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: TCMinpKD
Record Dates: First submitted 2023-02-26; First posted 2023-03-08 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Proteinuria; Kidney Diseases; Hereditary Nephropathy
Keywords: Traditional Chinese Medicine; anti-proteinuric
MeSH Terms: conditions — Proteinuria; Kidney Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): TCM+Routine therapy are used first for 12 weeks, followed by 2 weeks wash-out period, then Routine therapy for 12 weeks.
  TCM as Gu Shen Juan Yu Formula: 3g or 6g or 12g each time based on weight (3g for W≤20kg, 6g for 20-30kg, or 12g for W>30kg), 2 times a day for 12 weeks, orally.
  The GSJYF samples were made and packed by Shanghai Fangxin Pharmaceutical Technology Co., LTD. with lot number of 20230830.
  Routine therapy: with stable dose of ACE inhibitors/ angiotensin II receptor blocker.
  Interventions: Drug: TCM+ Routine Therapy; Drug: Routine Therapy
- Group B (Experimental): Routine therapy are used first for 12 weeks, followed by 2 weeks wash-out period, then TCM+Routine therapy for 12 weeks.
  TCM as Gu Shen Juan Yu Formula: 3g or 6g or 12g each time based on weight (3g for W≤20kg, 6g for 20-30kg, or 12g for W>30kg), 2 times a day for 12 weeks, orally.
  The GSJYF samples were made and packed by Shanghai Fangxin Pharmaceutical Technology Co., LTD. with lot number of 20230830.
  Routine therapy: with stable dose of ACE inhibitors/ angiotensin II receptor blocker.
  Interventions: Drug: TCM+ Routine Therapy; Drug: Routine Therapy

INTERVENTIONS:
Drug: TCM+ Routine Therapy — The Gu Shen Juan Yu Formula contains 11 herbs and it is available in liquid form for patients. Patients will receive Gu Shen Juan Yu Formula, 3g or 6g or 12g each time based on weight (3g for W≤20kg, 6g for 20-30kg, or 12g for W>30kg), 2 times a day for 12 weeks, orally.
  Routine therapy: Patients receiving a stable dose of ACEI/ARB will be continued.
  Other Names: Gushen Juanyu Formula+ACEI/ARB
Drug: Routine Therapy — Patients receive a stable dose of ACEI/ARB drug as a routine therapy.
  Other Names: ACEI/ARB

SUMMARY:
The purpose of this study is to determine whether traditional Chinese medicine, Gu Shen Juan Yu Formula, as complementary treatment is safe and effective in the treatment of Inherited Proteinuric Kidney Disease.

DETAILED DESCRIPTION:
Current therapy for inherited proteinuric kidney disease remains limited. Renin-angiotensin-aldosterone-system (RAAS) inhibitors such as Angiotensin converting enzyme inhibitors (ACEI) or angiotensin II receptor blockers (ARBs) help to control proteinuria and slow the progression of kidney function loss. However, a substantial proportion of patients progress to end-stage renal disease, which is partly associated with high residual proteinuria. Novel therapies to decrease proteinuria and limit CKD progression are needed. Traditional Chinese medicine (TCM) has been extensively used in China for thousands of years and favored in treatment of chronic disease for multi-factorial, multi-target action.

The investigators' hypothesis is that this traditional Chinese medicine, targeted to podocyte injury and repair named Gu Shen Juan Yu Formula, can significantly reduce proteinuria and delay renal function loss in patients with proteinuric kidney disease. To test this hypothesis, the investigators plan to initiate a multicenter, open-label, two-arm, crossover, randomized clinical trial in 72 children with proteinuria kidney disease. The study population will consist of children with proteinuria who are on receiving routine therapy such as ACE inhibitor or angiotensin II receptor blocker treatment. In this study, participants were randomly assigned (1:1) to receive first either TCM+Routine Therapy or Routine Therapy for 12 weeks. A 2 weeks washout period was used before crossover.

The primary objective was to measure the change of urine protein excretion and estimated glomerular filtration rate (eGFR) during the treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Aged 3-18 years；
* Proteinuria associated with hereditary nephropathy, which was confirmed by mutations in podocyte genes or syndromal genes (including collagens);
* Urine protein more than 500 mg/24 hours and/or UPCR (in first-morning void) more than 0.5 mg/mg at time of baseline despite ACEI or ARB treatment for at least 3 months;
* Estimated GFR ≥ 45 ml/min/1.73m2 (estimated with Schwartz formula);
* Without any immunosuppressive medications such as corticosteroids, calcineurin inhibitors, etc；
* On a stable dose of ACEI or ARB for at least 4 weeks；
* Willingness to give written consent and comply with the study protocol.

Exclusion Criteria:

* Diagnosed with Nephronophthisis, Polycystic kidney disease etc;
* With abnormal liver function, ALT or AST >3.0 x upper limit of normal (ULN) at enrollment;
* Receiving immunosuppressive therapy (including corticosteroids, and other immune suppressive medicine) within three months prior to enrollment;
* Receiving other traditional Chinese medicine and/or its analogue which can reduce proteinuria within the past 2 weeks. Patients who are taking other TCM treatment could be enrolled after 2 weeks of wash out period;
* Has undergone major organ transplantation (e.g. heart, kidney, liver);
* Any medication, surgical or medical condition which might significantly alter the absorption, distribution, or metabolism including, but not limited to any of the following: active inflammatory bowel disease, received major gastrointestinal tract surgery;
* History of noncompliance to medical regimens or inability to comply with the study and follow-up procedures.

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 72 (Actual)
Dates: Start 2023-09-17 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Percentage change in urinary protein-creatinine ratio (UPCR) from baseline to week 26 | baseline, week 12, week 14, week 26
  UPCR in first-morning spot urine samples are measured at baseline, week 12, week 14, and week 26. It is a repeated measurement.
Changes in estimated glomerular filtration rate (eGFR) from baseline to week 26 | baseline, week 12, week 14, week 26
  eGFR will be evaluated using Schwartz formula (eGFR=k*height(cm)/serum creatinine(umol/L)), k=36.5). Serum creatinine are measured at baseline, week 12, week 14, week 26. Serum creatinine is a repeated measurement.
Percentage change in urinary albumin-creatinine ratio (UACR) from baseline to week 26 | baseline, week 12, week 14, week 26
  UACR in first-morning spot urine samples are measured at baseline, week 12, week 14, and week 26. UPCR is a repeated measurement.
Percentage change in 24-hour protein from baseline to week 26 | baseline, week 12, week 14, week 26
  24-hour urine samples are measured at baseline, week 12, week 14, and week 26. 24-hour proteinuria is a repeated measurement.

SECONDARY OUTCOMES:
Changes in serum albumin from baseline to week 26 | baseline, week 12, week 14, week 26
  Serum albumin are measured at baseline, week 12, week 14, and week 26. Serum albumin is a repeated measurement.
Changes of Traditional Chinese Medicine syndrome scores after treatment | Baseline, week 26
  A TCM syndrome scale points are used to evaluate the Traditional Chinese Medicine syndromes at baseline, and week 26. The minimum values is 0 and maximum values is 36. The higher scores mean a severe status.
Changes in liver function parameters from baseline to week 26: Alanine Aminotransferase (ALT) | baseline, week 12, week 14, week 26
  Blood samples are measured at baseline, week 12, week 14, week 26 to evaluate ALT
Changes in liver function parameters from baseline to week 26: Aspartate Aminotransferase (AST) | baseline, week 12, week 14, week 26
  Blood samples are measured at baseline, week 12, week 14, week 26 to evaluate AST

OTHER OUTCOMES:
Number of subjects reporting adverse events （AEs）during the treatment period | baseline to week 26
  Number of subjects with AEs as a measure of safety

CONTACTS AND LOCATIONS:
Overall Officials: Hong Xu, PhD, Study Chair — Children's Hospital of Fudan University
Locations (9):
- China (9):
  - Anhui Provincial Children's Hospital, Hefei, Anhui
  - First Affiliated Hospital, Sun Yat-Sen University, Guangzhou, Guangzhou
  - Children's Hospital Affiliated to Zhengzhou University/Henan Children's Hospital, Zhengzhou, Henan
  - Wuhan Children's Hospital,Tongji Medical College, Huazhong University of Science and Technology., Wuhan, Hubei
  - Children's Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - Shandong Provincal Hospital, Shandong, Shandong
  - The Children's Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Children's Hospital of Fudan University, Shanghai
  - Xuzhou Children's Hospital, Xuzhou

IPD SHARING:
Plan to Share IPD: No